CLINICAL TRIAL: NCT05490134
Title: Evaluating the Specific Role of Endogenous Opioids as the Mechanism Underlying tAN-based Analgesia in Healthy Individuals
Brief Title: RM1 Project 1 - tAN Naloxone
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Jeffrey Borckardt, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00122762
Record Dates: First submitted 2022-08-02; First posted 2022-08-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Naloxone; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: All participants will be randomized to one of four stimulation groups in a 1:1:1:1 fashion such that each group will have 34 participants. Within each group, participants will be randomized to either receive naloxone or saline on their first visit, and the opposite on their second visit. The drug visit will be counterbalanced within each group to avoid a potential order confound.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ABVN Only Stimulation (Experimental): 30 minutes of ABVN Only stimulation (15Hz stimulation of cymba conchae).
  Interventions: Drug: Naloxone; Drug: Saline
- ATN Only Stimulation (Experimental): 30 minutes of ATNS Only stimulation (100Hz stimulation adjacently anterior to the tragus)
  Interventions: Drug: Naloxone; Drug: Saline
- Combination (ABVN + ATN) Stimulation (Experimental): 30 minutes of Combo stimulation (stimulation of both the 15Hz cymba conchae and 100HZ adjacently anterior to the tragus)
  Interventions: Drug: Naloxone; Drug: Saline
- Sham Stimulation (Experimental): 30 minutes of Sham (15Hz stimulation of the earlobe)
  Interventions: Drug: Naloxone; Drug: Saline

INTERVENTIONS:
Drug: Naloxone — A 0.15 mg/kg bolus dose of naloxone in 10ml normal saline will be administered via an intravenous (IV) line inserted into the antecubital vein of the non-dominant arm.
Drug: Saline — 0.15mg/kg bolus of normal saline in 10ml normal saline will be administered via an intravenous (IV) line inserted into the antecubital vein of the non-dominant arm.
  Other Names: Placebo

SUMMARY:
This two-visit, randomized, double-blind, sham-controlled trial, uses a novel naloxone blockade model in 136 individuals to determine whether the analgesic effects of a 30-minute transcutaneous auricular neurostimulation (tAN) intervention are mediated through a release of endogenous opioids. Analgesic effects of four various stimulation interventions will be measured (auricular vagus, auricular trigeminal, combination, or sham) while varying the type of intravenous (IV) infusion (either naloxone or saline) a participant is administered to determine whether the analgesic effects are mitigated by pharmacological opioid receptor blockade.

DETAILED DESCRIPTION:
The demand for chronic pain treatment has demonstrated an unprecedented increase over the last several decades, in part contributing to an unsustainable surge in opioid prescriptions. Countless patients were escalated to prolonged, high-dose opioid regimens over years of treatment. By 2014, 5.4% of US adults were estimated to use prescription opioids on a long-term basis. As the harms of opioid proliferation became increasingly clear, a dramatic paradigm shift occurred in which these drugs came to be seen as often more dangerous than beneficial for chronic pain. New clinical guidelines highlighted the risks of high-dose regimens as well as limited benefits, particularly insufficient analgesia, associated with long-term use. According to this new perspective, the preferred therapeutic modality for many patients is to significantly reduce, or even completely stop, using opioids.

Stimulation of the auricular branch of the vagus nerve (ABVN) has demonstrated additional benefits for reducing the need for opioids for pain as well as lessening opioid withdrawal symptoms. Clinical trials of ABVN stimulation as an adjunctive treatment for pain have noted decreased intake of tramadol, remifentanil, morphine, as well as naproxen plus tramadol. A pioneering study of electrical stimulation at the cymba conchae in eight persons with opioid use disorder found significantly reduced withdrawal symptoms: first, decreases in anxiety, craving for opioids, chills, nausea; second, reduced bone and joint pain. Results in follow-up clinical trials bolstered the efficacy of ABVN stimulation for opioid withdrawal. More recently, an open-label trial of simultaneous ABVN and trigeminal stimulation found reduced withdrawal symptoms and decreased need for morphine maintenance in newborns with neonatal opioid withdrawal syndrome (see Preliminary Studies, below). This method of simultaneous vagal and trigeminal stimulation via the external ear is known as transcutaneous auricular neurostimulation (tAN), as the targets of electrical stimulation include the ABVN and auriculotemporal nerve (ATN), which is a branch of the mandibular division of the trigeminal nerve. Electrodes applied to select dermatome regions can target ear neural structures and deliver non-invasive VNS and TNS.

Use of tAN devices for pain relief is an attractive alternative to pharmacologic and opioid-based approaches because it is safe and effective and presents no addiction liability. In order to increase clinical adoption and optimize efficacy of these devices, the mechanism of action must be fully characterized.

This study is investigating the anti-pain mechanism behind tAN in a healthy cohort. This study begins to understand whether the anti-pain effects are driven by a release of endogenous opioids - and will accomplish this by administering tAN during aμ-opioid receptor blockade (via naloxone IV). Administering tAN concurrently with IV Naloxone or Saline (control) will allow us to better understand what underlying mechanism drives the analgesic effects of tAN, and whether the blockade of opioid receptors blocks the anti-pain effects of tAN.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Have the capacity and ability to provide one's own consent and sign the informed consent document

Exclusion Criteria:

* Contraindicated for MRI.
* Any current or recent untreated medical, neurological, or psychiatric conditions
* Metal implant devices in the head, heart or neck.
* History of brain surgery.
* History of myocardial infarction or arrhythmia, bradycardia.
* Personal or family history of seizure or epilepsy or personal use of medications that substantially reduce seizure threshold (e.g., olanzapine, chlorpromazine, lithium).
* Personal history of head injury, concussion, or self-report of moderate to severe traumatic brain injury.
* Individuals suffering from frequent/severe headaches.
* Individuals with a reported history of psychosis or mania, or individuals who are actively manic or psychotic.
* Regular or recent pain medication use
* Moderate to severe alcohol or substance use disorder.
* Psychotropic or cardiac medicines that may interact with naloxone
* Positive urine drug screen for opiate use
* Females who are pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Thermal Pain Thresholds | Change from Baseline Pain Threshold at Post-Stimulation Timepoint
  Using a quantitative sensory testing paradigm, the investigators will systematically determine information on thermal pain tolerance thresholds (degrees celsius) using a 30 × 30 mm thermode attached to the left forearm of participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No